CLINICAL TRIAL: NCT00487643
Title: Normal Lacritin Levels in Human Tears- Development of a New Clinical Assay
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: University of Virginia (Other); James Madison University (Other); Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Samantha B. Rodgers, MD, Assistant Director, Warfighter Refractive Eye Surgery Program and Research Center at FT Belvoir, Fort Belvoir Community Hospital
Other Study IDs: WRAMC WU# 07-23021
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Tear Protein Lacritin in Human Tears
Keywords: Lacritin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Tear Collection — The tear sample will be collected from the left eye of each subject. Subjects wearing contact lenses will be instructed to remove their lenses and wait at least 5 minutes before proceeding with the tear collection procedure. The patient will then be instructed to sit with eyes gently closed for two minutes after instilling one (1) drop of 0.5% proparacaine on the cornea and conjunctiva. Tear collection was accomplished by using a polyester fiber rod wick. This wick will be placed in contact with the tear fluid at the lower cul-de-sac for a minimum time to obtain fluid without irritating the subject's eye approx. for 3 to 5 minutes.

SUMMARY:
Purpose: to build a library of normal tear lacritin values by collecting tears from normal adult human subjects and to develop a non-invasive clinical assay for lacritin. Such an assay will provide more sensitive indicators of eye disease for clinicians and determine if a particular therapy, such as recombinant lacritin drops, is of benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Military health care beneficiary between the ages of 21-55.
2. Male or female, of any race, and at least 21 years old and not older than 55 years old at the time of tear collection.
3. Appropriately aged individuals who report that their eyes are "normal" and who have no active eye illness as determined by principal investigator or sub-investigator.
4. Ability and willingness to understand and provide informed consent to participate in this study.

Exclusion Criteria:

1. Irritated eye reflected by patient statements or finding of "red" eye.
2. Individuals with any infections or inflammatory ocular condition (e.g. have "pink eye" or uveitis).
3. Individuals diagnosed with dry eye or other ocular surface condition, including but not restricted to neurotrophic keratitis, anterior basement membrane dystrophy, and recurrent corneal erosions.
4. Individuals who are on any topical eye medications.
5. Anyone who reports previous reaction or the possibility of an allergic reaction to 0.5% proparacaine.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Military health care beneficiary between the ages of 21-55.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
lacritin levels in human tears | 2 minutes after instilling anesthetic eyedrop

CONTACTS AND LOCATIONS:
Overall Officials: Kraig S. Bower, MD, Principal Investigator — WRAMC
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States